CLINICAL TRIAL: NCT02441036
Title: Evaluation of Changes in Gene Expression Following Ultherapy® Treatment
Brief Title: Gene Expression Following Ultherapy® Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to non-safety reasons
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ULT-140
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-12

CONDITIONS: Skin Laxity
Keywords: Gene expression and protein production
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (5):
- Group 1 - 1-3 hours prior (Active Comparator): Subjects will receive Ultherapy treatment 1-3 hours prior to tissue resection.
  Interventions: Device: Ultherapy Treatment
- Group 2 - 1 day prior (Active Comparator): Subjects will receive Ultherapy treatment 1 day prior to tissue resection.
  Interventions: Device: Ultherapy Treatment
- Group 3 - 3 days prior (Active Comparator): Subjects will receive Ultherapy treatment 3 days prior to tissue resection.
  Interventions: Device: Ultherapy Treatment
- Group 4 - 7 days prior (Active Comparator): Subjects will receive Ultherapy treatment 7 days prior to tissue resection.
  Interventions: Device: Ultherapy Treatment
- Group 5 - 45 days prior (Active Comparator): Subjects will receive Ultherapy treatment 45 days prior to tissue resection.
  Interventions: Device: Ultherapy Treatment

INTERVENTIONS:
Device: Ultherapy Treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ulthera System Treatment

SUMMARY:
Up to 25 subjects will be enrolled and randomized. Randomized subjects will receive one single-side Ulthera® treatment in the pre-auricular region on the face. At each subject's scheduled facelift procedure, resected tissue will be obtained for analysis.

DETAILED DESCRIPTION:
This is a prospective, multi-center, pilot clinical trial to evaluate the molecular changes following an Ultherapy® treatment. Subjects will be randomized to one of five treatment groups and, based on study group assignment, will receive one single-side Ultherapy® treatment at varying timepoints prior to an already planned facelift procedure. Treatment will be delivered to the pre-auricular region on one side of the face; the contralateral side will serve as control. During an already planned facelift procedure, treated and non-treated resected tissue will be obtained for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 45 to 70 years.
* Subject in good health.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control during the study.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other Non-Steroidal Anti-Inflammatory Drug (NSAID) prior to study treatment and chronic use during the entire post-treatment study period.
* Willingness and ability to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Significant scarring in the area(s) to be treated that would interfere with assessing results.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included.)
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within four weeks prior to study participation or during the study.
* Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* BMI equal to or greater than 30.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
* History of the following cosmetic treatments in the area(s) to be treated:

  1. Skin tightening procedure within the past year;
  2. Injectable filler of any type within the past:

  i. 12 months for Hyaluronic acid fillers (e.g. Restylane)

ii. 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)

iii. 24 months for Long-lasting Hyaluronic acid (Juvéderm Voluma) and Poly-L-Lactic acid fillers (e.g. Sculptra)

iv. Ever for permanent fillers (e.g. Silicone, ArteFill)

c. Neurotoxins within the past three months;

d. Ablative resurfacing laser treatment within the past six months;

e. Nonablative, rejuvenative laser or light treatment within the past six months;

f. Surgical dermabrasion or deep facial peels; or

g. Facelifts within the past year.

* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Topical Retinoids within the past two weeks;
  3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
  4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Ulthera, Inc
Locations (2):
- United States (2):
  - North Valley Plastic Surgery, Phoenix, Arizona
  - Campbell Facial Plastic Surgery, Mequon, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-3 Hours Before Resection: Subjects will receive Ultherapy treatment 1-3 hours prior to tissue resection
- 1 Day Before Resection: Subjects will receive Ultherapy treatment 1 day prior to tissue resection
- 3 Days Before Resection: Subjects will receive Ultherapy treatment 3 days prior to tissue resection
- 7 Days Before Resection: Subjects will receive Ultherapy treatment 7 days prior to tissue resection
- 45 Days Before Resection: Subjects will receive Ultherapy treatment 45 days prior to tissue resection
Period: Overall Study
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
Started | 3 | 5 | 3 | 4 | 1
Treated | 3 | 5 | 3 | 4 | 1
Tissue Resected | 3 | 4 | 3 | 3 | 1
Completed | 3 | 4 | 3 | 3 | 1
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — No tissue resected | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection | Total
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 1 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 1 | 3 | 1 | 12
  >=65 years | 0 | 1 | 2 | 1 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [48.7 to 56.6] | 58.9 [50.0 to 68.8] | 65.3 [59.3 to 69.5] | 60.0 [52.1 to 66.8] | 63.3 [63.3 to 63.3] | 59.3 [48.7 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 1 | 15
  Male | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 3 | 4 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gene Expression in Facial Skin Tissue Treated With Ultherapy Compared to Control (Untreated) Tissue Through Microarray Profiling
Description: RNA will be extracted from treated and untreated (control) tissue samples obtained from 15 study subjects. For each subject tissue of the contra-lateral side of the face served as a control and will not receive Ultherapy treatment.
  OneArray Human Gene Expression microarray will be used for microarray profiling. Clustering Analysis will be performed to identify differences between treated vs. control samples and the up and down-regulated genes will be represented in a heatmap. The number of differentially expressed genes in treated samples compared to control samples will be determined for every study group.
Time Frame: 1-3 hours to up to 45 days following Ultherapy treatment
Population: Unanticipated sample collection/preservation issues reduced the number of samples available to 9 samples out of the 15 minimum required. These did not represent all intended time points. Study analyses were not performed as achieving meaningful outcomes was not possible with the small sample of specimens, i.e., data were not collected.
Groups:
- 45 Days Before Resection: Subjects will receive Ultherapy treatment 45 days prior to tissue resect
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Changes in Gene Expression of Apoptotic Genes Induced in Tissues Treated With Ultherapy Relative to Control (Untreated) Tissues by PCR Array
Description: Real-time PCR array will be performed to assess differences in gene expression of a cluster of 84 genes related to apoptosis (e.g. Annexin V, Caspacin, TNF ligands and their receptors, members of the bcl-2, caspase, IAP, TRAF, CARD, death domain, death effector domain, and CIDE families, as well as genes involved in the p53 and DNA damage pathways) between control versus treated tissues. The number of differentially expressed genes in treated samples compared to control samples will be determined for every study group.
Time Frame: 1-3 hours to up to 45 days following Ultherapy treatment
Population: as for outcome 1
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Changes in Gene Expression of Heat Shock Proteins Genes Induced in Tissues Treated With Ultherapy Relative to Control (Untreated) Tissues by PCR Array
Description: Real-time PCR array will be performed to assess differences in gene expression of a cluster of 84 Heat Shock Protein genes that regulate protein folding (e.g. HSP90 (81 to 99 kD), HSP70 (65 to 80 kD), HSP60 (55 to 64 kD), HSP40 (35 to 54 kD), small HSPs (=34 kD) and other chaperone cofactors) between control versus treated tissues. The number of differentially expressed genes in treated samples compared to control samples will be determined for every study group.
Time Frame: 1-3 hours to up to 45 days following Ultherapy treatment
Population: as for outcome 1
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Changes in Protein Expression in Tissues Treated With Ultherapy Compared to Control (Untreated) Tissue by Immunohistochemistry
Description: Protein expression of apoptotic genes and heat shock proteins of interest identified in the three previous outcomes will be analyzed. Embedded or frozen section tissues will be stained for specific proteins previously identified. The number of subjects with differentially expressed proteins in treated samples compared to control samples will be determined for every study group.
Time Frame: 1-3 hours to up to 45 days following Ultherapy treatment
Population: as for outcome 1
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed for up to 45 days post-treatment or until event resolution.
Arm/Group | 1-3 Hours Before Resection | 1 Day Before Resection | 3 Days Before Resection | 7 Days Before Resection | 45 Days Before Resection
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No